CLINICAL TRIAL: NCT03802929
Title: The DOMESTIC Study: Diagnostic and Prognostic Prediction Models for Patients With Venous Thromboembolism in China
Brief Title: Diagnostic and Prognostic Prediction Models for Chinese Patients With Venous Thromboembolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ya-Wei Xu (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Head of Cardiology, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: DOMESTIC
Record Dates: First submitted 2018-12-26; First posted 2019-01-14 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood collected at various time points according to the study cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Cohort: Derivation Cohort of Diagnostic Prediction Model:
  Participants will be recruited from the emergency department of five general urban hospitals in China, including Shanghai Tenth People's Hospital; Nanfang Hospital of Southern Medical University; First Affiliated Hospital, Sun Yat-Sen University; Zhongshan Hospital Xuhui Branch, Fudan University; Shanghai Baoshan Luo Dian Hospital; from March 1, 2019. The investigators will randomly assign 70% participants to a derivation cohort.
  Derivation Cohort of Prognostic Prediction Model:
  Patients with VTE from 5 thrombosis centers in China, including Shanghai Tenth People's Hospital; Nanfang Hospital of Southern Medical University; First Affiliated Hospital, Sun Yat-Sen University; Zhongshan Hospital Xuhui Branch, Fudan University; Shanghai Baoshan Luo Dian Hospital; between January 2014 and December 2018.
- Validation Cohort: Validation Cohort of Diagnostic Prediction Model:
  The investigators plan to randomly assign 30% participants for developing the diagnostic prediction model to a Validation cohort.
  Validation Cohort of Prognostic Prediction Model:
  New individuals selected by the same inclusion and exclusion criteria as the derivation cohort of prognostic prediction model from the same institutions as a validation cohort of prognostic prediction model will be recruited from January 2019.

SUMMARY:
The objective of this proposal is to develop and validate diagnostic and prognostic (including short-term and long-term prognoses) prediction models for patients with venous thromboembolism (VTE) in China.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), which clinically manifests as deep vein thrombosis (DVT) and pulmonary embolism (PE), is one of the leading causes of mortality that need to be accurately diagnosed and effectively managed. Although a number of clinical decision rules in the domain of VTE have been presented in the literature, such as the well-known prediction models developed by Wells and colleagues, the prognostic models to assess VTE recurrence risk in patients who suffered from a VTE or the Pulmonary Embolism Severity Index (PESI) for short-term mortality risk in PE patients, and various other diagnostic models for both DVT and PE. They are few designed for Chinese patients. The primary objective of this proposal is to develop and validate diagnostic and prognostic (including short-term and long-term prognoses) prediction models for patients with VTE in China.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old
2. First episode of PE and/or DVT (diagnosed by pulmonary angiogram, chest computed tomography pulmonary angiography(CTPA), Ventilation/Perfusion (V/Q) lung scan read as high probability by the radiologist, and/or (+) bilateral lower limb venous compression ultrasonography (CCUS))

Exclusion Criteria:

1. Patients with prior VTE
2. Cannot provide written informed consent
3. Unable to read questionnaire in Chinese or English
4. a record of pregnancy in the preceding 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Development and validation of diagnostic prediction model:
  Participants will undergo recruitment from the emergency department of five general urban hospitals in China, including Shanghai Tenth People's Hospital; Nanfang Hospital of Southern Medical University; First Affiliated Hospital, Sun Yat-Sen University; Zhongshan Hospital Xuhui Branch, Fudan University; Shanghai Baoshan Luo Dian Hospital; from March 1, 2019.
  Development and validation of prognostic prediction model:
  The investigators will identify patients with VTE from 5 thrombosis centers in China, including Shanghai Tenth People's Hospital; Nanfang Hospital of Southern Medical University; First Affiliated Hospital, Sun Yat-Sen University; Zhongshan Hospital Xuhui Branch, Fudan University; Shanghai Baoshan Luo Dian Hospital; between January 2014 and December 2018 using the Hospital Information Manage System(HIMS) database.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Death from all causes | 5-year
  Death from all causes during follow-up
Death from all causes | 30-day
  Death from all causes during hospitalization

SECONDARY OUTCOMES:
Number of Participants with Recurrent VTE | 5-year
  Recurrent symptomatic DVT confirmed by venography or color duplex sonography or recurrent symptomatic pulmonary embolism confirmed by ventilation-perfusion scanning, CTPA, or pulmonary angiogram.
Number of Participants with Chronic Thromboembolic Pulmonary Hypertension(CTEPH) | 5-year
  CTEPH can be diagnosed by an echocardiogram or a CTPA.

OTHER OUTCOMES:
Number of Participants with Cardiogenic Shock | 30-day
  Cardiogenic shock defined as hemodynamic instability(systolic blood pressure<90 mm Hg, or use of inotropic support）

CONTACTS AND LOCATIONS:
Overall Officials: Dachun Xu, Ph.D, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang F, Wang L, Yan C, Chang X, Wang H, Zhu K, Xu Y, Xu D. Algorithms of Electrocardiographic Changes for Quantitative and Localization Analysis of Thrombus Burden in Patients with Acute Pulmonary Thromboembolism. Rev Cardiovasc Med. 2023 Oct 7;24(10):281. doi: 10.31083/j.rcm2410281. eCollection 2023 Oct. PMID 39077587